CLINICAL TRIAL: NCT01058057
Title: Atorvastatin Pre-Treatment Influences the Risk of Percutaneous Coronary Intervention Study 2
Brief Title: Atorvastatin Pre-Treatment Influences the Risk of Percutaneous Coronary Intervention (PCI) Study 2
Acronym: TIPS-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Prof. Anna Sediva, MD, PhD, University Hospital Motol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC EK-150/08
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease; Coronary Angioplasty
Keywords: atorvastatin; percutaneous coronary intervention; periprocedural myocardial infarction; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental): Atorvastatin 80mg seven days pre-treatment before PCI
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — atorvastatin 80mg p.o. daily seven days before PCI
  Other Names: Torvacard

SUMMARY:
This study investigates potential protective effect of atorvastatin pre-treatment in patient with stable coronary artery disease undergoing percutaneous coronary intervention (PCI) on chronic statin therapy. Patients are randomized into two groups: atorvastatin pre-treatment group (80mg atorvastatin seven days before PCI) and control group (PCI without atorvastatin pretreatment, chronic statin treatment). Endpoint is myocardial infarction measured by troponin I and creatine kinase myocardial band.

DETAILED DESCRIPTION:
This randomized study investigates potential protective effect of high dose atorvastatin pre-treatment in patient with stable coronary artery disease undergoing percutaneous coronary intervention (PCI) and chronic statin therapy.

Two arms:

1. atorvastatin pre-treatment group (80mg atorvastatin for seven days)
2. control group (without atorvastatin pre-treatment, chronic statin treatment)

Primary endpoint:

Periprocedural myocardial infarction measured by troponin I level (time frame 24 hours)

Secondary endpoint:

Periprocedural myocardial infarction measured by creatine kinase myocardial band (time frame 24 hours)

ELIGIBILITY:
Inclusion Criteria:

* Indication for percutaneous coronary intervention
* Informed consent
* Chronic statin therapy

Exclusion Criteria:

* Acute coronary syndrome in last 14 days
* Renal insufficiency (creatinine more 150 umol/l)
* Diseases severely limiting prognosis
* Previous participation in this study
* Chronic occlusion of the coronary artery, bypass intervention, left main intervention
* Chronic statin treatment with atorvastatin 80mg daily and rosuvastatin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
periprocedural myocardial infarction measured by troponin I level | 24 hours after PCI

SECONDARY OUTCOMES:
periprocedural myocardial infarction measured by creatinine kinase myocardial band | 24 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: David Zemanek, MD, Principal Investigator — Department of Cardiology, University Hospital Motol; Josef Veselka, Prof., MD., PhD., Study Chair — Department of Carldiology, University Hospital Motol
Locations (1):
- Dpt. of Cardiology, University Hospital Motol, Prague, Czechia

REFERENCES:
- [Background] Veselka J, Zemanek D, Hajek P, Maly M, Adlova R, Martinkovicova L, Tesar D. Effect of two-day atorvastatin pretreatment on the incidence of periprocedural myocardial infarction following elective percutaneous coronary intervention: a single-center, prospective, and randomized study. Am J Cardiol. 2009 Sep 1;104(5):630-3. doi: 10.1016/j.amjcard.2009.04.048. Epub 2009 Jun 24. PMID 19699335
- [Background] Di Sciascio G, Patti G, Pasceri V, Gaspardone A, Colonna G, Montinaro A. Efficacy of atorvastatin reload in patients on chronic statin therapy undergoing percutaneous coronary intervention: results of the ARMYDA-RECAPTURE (Atorvastatin for Reduction of Myocardial Damage During Angioplasty) Randomized Trial. J Am Coll Cardiol. 2009 Aug 4;54(6):558-65. doi: 10.1016/j.jacc.2009.05.028. Epub 2009 Jul 2. PMID 19643320
- [Background] Mood GR, Bavry AA, Roukoz H, Bhatt DL. Meta-analysis of the role of statin therapy in reducing myocardial infarction following elective percutaneous coronary intervention. Am J Cardiol. 2007 Sep 15;100(6):919-23. doi: 10.1016/j.amjcard.2007.04.022. Epub 2007 Jun 26. PMID 17826370